CLINICAL TRIAL: NCT01830920
Title: A Multi-Center, Parallel-Group, Randomized, Double Blind, Adaptive Study Investigating the Safety and Efficacy of THR-184 in Patients at Increased Risk of Developing Cardiac Surgery Associated-Acute Kidney Injury (CSA-AKI)
Brief Title: A Study of THR-184 in Patients at Risk of Developing Cardiac Surgery Associated-Acute Kidney Injury (CSA-AKI)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thrasos Innovation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A-003; 2741202 (Other: CTI Clinical Trial and Consulting Services, Inc.)
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; AKI; Cardiac surgery
MeSH Terms: conditions — Acute Kidney Injury | interventions — THR-184; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): An identical appearing placebo will be administered.
  Interventions: Drug: Placebo
- THR-184 Dose 1 (Experimental): THR-184 initial pre-surgery low dose followed by (3) post surgery doses at the low dose.
  Interventions: Drug: THR-184
- THR-184 Dose 2 (Experimental): THR-184 initial pre-surgery mid-dose followed by (3) post surgery doses at the low dose.
  Interventions: Drug: THR-184
- THR-184 Dose 3 (Experimental): THR-184 initial pre-surgery high dose followed by (3) post surgery doses at the low dose.
  Interventions: Drug: THR-184
- THR-184 Dose 4 (Experimental): THR-184 initial pre-surgery high dose followed by (3) post surgery doses ~80% of the pre-surgery dose.
  Interventions: Drug: THR-184

INTERVENTIONS:
Drug: THR-184 — THR-184 is a synthetic oligopeptide administered intravenously.
  Other Names: Synthetic oligopeptide
  Arms: THR-184 Dose 1; THR-184 Dose 2; THR-184 Dose 3; THR-184 Dose 4
Drug: Placebo — A normal saline solution identical in appearance to the active drug solution
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether THR-184 when administered around the time of cardiac surgery that requires cardiopulmonary bypass can prevent or ameliorate the development of acute kidney injury.

DETAILED DESCRIPTION:
The study has been designed to include patients scheduled for cardiac surgery who are considered at increased risk for developing CSA-AKI. The eligibility criteria are intended to enrich the study population with such patients.

Stage 1 consisted of 140 patients randomized in a 1:1:1:1 ratio (approximately 35 patients per treatment arm) to Placebo or to one of three (3) THR-184 dose arms:

* initial pre-surgery low dose of THR-184 by three (3) post-surgery doses at the low dose, or
* initial pre-surgery middle dose of THR-184 followed by three (3) post-surgery doses at the low dose, or
* initial pre-surgery high dose of THR-184 followed by three (3) post-surgery doses at the low dose

An interim analysis (IA) was performed by the Independent Statistical Center (ISC) and presented to the Independent Data Monitoring Committee (IDMC). The IDMC indicated no safety concerns and recommended that the study continue with the placebo arm and the initial pre-surgery high dose arm. Additionally, another dosing arm will be added, which will increase the dose post-surgery.

Stage 2 will consist of approximately 270 patients randomized in a 1:1:2 ratio to Placebo or to a dose selected from one of the two (2) THR-184 dose arms:

* initial pre-surgery high dose of THR-184, followed by (3) post-surgery doses at the original low dose;
* initial pre-surgery high dose of THR-184, followed by (3) post-surgery doses at ~80% of the pre-surgery dose

Study treatment (THR-184 or placebo) will consist of one 60-minute IV infusion administered prior to surgery, followed by a 60-minute IV infusion administered, beginning in the early post-operative period, and followed by two (2) additional 60-minute IV infusions administered, on consecutive days post-cardiac surgery.

The primary endpoint for the evaluation of efficacy in patients receiving THR-184, as compared to patients receiving Placebo, will be the proportion of patients developing CSA-AKI as measured by the Kidney Disease Improving Global Outcomes (KDIGO) criteria, as follows:

* Increase in Serum creatinine (SCr) by ≥0.3 mg/dl (>26.5 µmol/l) within 48 hours post-surgery; or
* Increase in SCr to ≥1.5 times a baseline which has been measured in the previous 7 days; or
* Urine volume <0.5 ml/kg/h for 6 hours post-operatively

If at least one of these measures is present by the 7 day assessment, a patient will be considered to have developed CSA-AKI.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and >18 years of age.
* Scheduled for a non-emergent coronary and/or valve surgery procedure requiring CPB, to include:

  * coronary artery bypass graft (CABG) alone;
  * aortic valve replacement or repair alone, with or without aortic root repair;
  * mitral, tricuspid, or pulmonic valve replacement or repair alone;
  * simultaneous replacement of several cardiac valves;
  * CABG with aortic, mitral, tricuspid, or pulmonic valve replacement or repair;
  * CABG with combined cardiac valve replacement or repair.
* Have the following risk factors for CSA-AKI:

  * eGFR ≥ 20 and < 30 ml/min/1.73m2 OR
  * eGFR ≥ 30 and < 60 ml/min/1.73m2 and ONE of the following additional risk factors (other than age ≥ 75 years) OR
  * eGFR ≥ 60 ml/min/1.73m2 and TWO of the following additional risk factors

Additional Risk Factors:

* Age ≥ 75 years;
* Combined valve & coronary surgery;
* Previous cardiac surgery with sternotomy;
* Documented NYHA Class III or IV within 1 year prior to surgery;
* Left ventricular ejection fraction (LVEF) ≤ 35% by invasive or noninvasive diagnostic cardiac imaging - echocardiography, nuclear imaging, computed tomography, magnetic resonance imaging or angiography performed within 90 days prior to surgery. (If LVEF ≤ 35% by any invasive or noninvasive imaging procedure, patient meets the risk factor.)
* Insulin-requiring diabetes;
* Non-insulin-requiring diabetes and the presence of ≥+2 proteinuria on urinalysis (medical history or dipstick);
* Preoperative anemia (hemoglobin <11g/dl for men and women).

Exclusion Criteria:

If any of the following criteria apply prior to surgery, the patient will be excluded from the study:

* Age > 85 years;
* Weight >174 kg or 383 lbs;
* The presence of AKI (KDIGO criteria) at the time of screening ;
* Surgery to be performed without CPB;
* Surgery to be performed under conditions of circulatory arrest or hypothermia with rectal temperature < 28°Celsius (82.4° Fahrenheit);
* eGFR (MDRD) <20 ml/min/1.73m2;
* Surgery for aortic dissection;
* Surgery to correct a major congenital heart defect (e.g., Tetralogy of Fallot, transposition of the great vessels, single ventricle, Ebsteins anomaly. Bicuspid aortic valve is not to be considered a congenital heart defect.);
* Prior organ transplantation;
* Dialysis-dependence;
* Administration of iodinated contrast media within 24 hours prior to cardiac surgery;
* If received contrast media prior to 24 hours and have AKI as defined by KDIGO criteria;
* Cardiogenic shock or haemodynamic instability within the 24 hours prior to surgery, including the anesthesia induction period; as defined by a systolic BP <80 mm Hg and pulse >120 beats per minute (bpm) and requirement for inotropes or vasopressors or other mechanical devices such as intra-aortic balloon counter-pulsation (IABP);
* Requirement for any of the following within seven (7) days prior to cardiac surgery:

  * defibrillator or permanent pacemaker,
  * mechanical ventilation,
  * intra-aortic balloon counter-pulsation (IABP),
  * left ventricular assist device (LVAD),
  * other forms of mechanical circulatory support (MCS);
* Cardiopulmonary resuscitation within 14 days prior to cardiac surgery;
* Known history of cancer within the past 5 years, except for carcinoma in situ of the cervix or adequately treated basal cell carcinoma of the skin;
* Known or suspected sepsis at time of screening;
* Known or suspected glomerulonephritis or interstitial nephritis at time of screening;
* Confirmed or treated endocarditis within previous 30 days prior to cardiac surgery;
* Other current active infection requiring antibiotic treatment;
* Patients with known active human immunodeficiency virus infection;
* Documented history of HIV antibodies;
* Patients with known active Hepatitis B (HBV) or Hepatitis C (HCV) infection;
* Documented history of HCV antibodies;
* Documented history of HBV antigens;
* Patients on immunosuppressant drugs or prednisone over the dose of 20 mg per day;
* Inadequate hepatic function, defined as total bilirubin or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 times the upper limit of normal (ULN) at time of screening or Child Pugh Class C liver disease ( see appendix 6) or higher;
* Any congenital coagulation disorder;
* Pregnancy or lactation;
* If patient has "Do Not Resuscitate" (DNR) status;
* Known hypersensitivity to the study drug or any of its excipients;
* Treatment with an investigational drug or participation in an interventional trial within 60 days prior to 1st dose of study drug;
* In the opinion of the investigator any disease processes or confounding variables that would inappropriately alter the outcome of the study;
* Inability to comply with the requirements of the study protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2013-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Orfanos, MBBCh, Study Director — Thrasos Innovation, Inc.
Locations (41):
- United States (31):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - Harbor - University of California Los Angeles Medical Center, Torrance, California
  - Danbury Hospital, Danbury, Connecticut
  - River City Clinical Research, Jacksonville, Florida
  - University of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Indiana Ohio Heart, Fort Wayne, Indiana
  - Indiana Heart-St. Vincent Medical Group, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - John Hopkins University, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - Covenant Medical Center, Saginaw, Michigan
  - Washington University, St Louis, Missouri
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - St. Peter's Hospital, Albany, New York
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Durham VA Medical Center, Durham, North Carolina
  - Lindner Research Center-Christ Hospital, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Erlanger Health System, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Soltero Cardiovascular Research Center, Dallas, Texas
  - University of Texas, Houston, Houston, Texas
  - Cardiothoracic Surgical Associates, Richmond, Virginia
- Canada (10):
  - Foothills Medical Centre, Calgary, Alberta
  - St-John Regional Hospital Facility, Saint John, New Brunswick
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut de Cardiologie de Montréal, Montreal, Quebec
  - Centre hospitalier de l'université de Montréal(CHUM)- Hôtel-Dieu, Montreal, Quebec
  - MUHC - Royal Victoria Hospital, Montreal, Quebec
  - Sacre Cœur Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | THR-184 Dose 1 | THR-184 Dose 2 | THR-184 Dose 3 | THR-184 Dose 4
Started | 126 | 46 | 48 | 125 | 107
Received Allocated Drug | 115 | 45 | 47 | 119 | 105
Completed | 105 | 40 | 40 | 109 | 99
Not Completed | 21 | 6 | 8 | 16 | 8
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 7 | 1
Not completed — Death | 3 | 3 | 5 | 4 | 4
Not completed — Other | 15 | 1 | 1 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | THR-184 Dose 1 | THR-184 Dose 2 | THR-184 Dose 3 | THR-184 Dose 4 | Total
Number analyzed (Participants) | 115 | 45 | 47 | 119 | 105 | 431
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 71.5 [65 to 80] | 68.8 [62 to 77] | 72.7 [66 to 79] | 72.5 [67 to 78] | 70.0 [64 to 77] | 71.3 [65 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 18 | 13 | 39 | 34 | 148
  Male | 71 | 27 | 34 | 80 | 71 | 283
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 2 | 5
  Asian | 2 | 2 | 0 | 1 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 1 | 5 | 3 | 17
  White | 105 | 40 | 44 | 110 | 95 | 394
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 1 | 2 | 2 | 7
Region of Enrollment [Number; unit: participants]
  Canada | 46 | 17 | 27 | 55 | 55 | 200
  United States | 69 | 28 | 20 | 64 | 50 | 231

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Kidney Injury (AKI)
Description: Acute kidney injury (AKI) is defined using the KDIGO criteria, in which AKI is defined as any of the following:
  * Increase in SCr by ≥0.3 mg/dl (≥26.5 µmol/l) within 48 hours; or
  * Increase in SCr to ≥1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
  * Urine volume <0.5 ml/kg/h for 6 hours.
Time Frame: 7 days
Population: Per Protocol Analysis set -
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | THR-184 Dose 1 | THR-184 Dose 2 | THR-184 Dose 3 | THR-184 Dose 4
Number analyzed (Participants) | 93 | 24 | 29 | 91 | 71
Participants | 73 | 18 | 22 | 71 | 50

2. Secondary Outcome: Incidence of AKI
Description: AKI is defined using the SCr-KDIGO criteria, defined as the following:
  * Increase in SCr by ≥0.3 mg/dl (≥26.5 µmol/l) within 48 hours; or
  * Increase in SCr to ≥1.5 times baseline, which is known or presumed to have occurred within the prior 7 days.
Time Frame: 7 days
Population: Per Protocol Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | THR-184 Dose 1 | THR-184 Dose 2 | THR-184 Dose 3 | THR-184 Dose 4
Number analyzed (Participants) | 93 | 24 | 29 | 91 | 71
Participants | 53 | 13 | 17 | 51 | 35

3. Secondary Outcome: Severity of AKI
Description: AKI is defined using the KDIGO criteria, in which AKI is defined as any of the following:
  * Increase in SCr by ≥0.3 mg/dl (≥26.5 µmol/l) within 48 hours; or
  * Increase in SCr to ≥1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
  * Urine volume <0.5 ml/kg/h for 6 hours.
  Staging of AKI is defined as the following:
  Stage 1: SCr 1.5 - 1.9 times baseline OR ≥0.3 mg/dL (≥26.5 µmol/L) increase, Urine output <0.5 ml/kg/hr for 6-12 hours Stage 2: SCr 2.0-2.9 times baseline, Urine output <0.5 ml/kg/h for ≥ 12 hours Stage 3: SCr 3.0 times baseline OR Increase in SCr to ≥5.0 mg/dL (≥353.6 µmol/L) OR Initiation of renal replacement therapy OR In patients <18 years, decrease in eGFR to <35 ml/min per 1.73 m^2, Urine output <0.3 ml/kg/h for ≥24 hours OR Anuria for ≥12 hours.
  No AKI is considered the best outcome, and Stage 3 the worst outcome.
Time Frame: 7 days
Population: Per Protocol Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | THR-184 Dose 1 | THR-184 Dose 2 | THR-184 Dose 3 | THR-184 Dose 4
Number analyzed (Participants) | 93 | 24 | 29 | 91 | 71
Participants
  No AKI | 20 | 6 | 7 | 20 | 21
  Stage I AKI | 47 | 10 | 12 | 48 | 29
  Stage II AKI | 23 | 7 | 9 | 22 | 18
  Stage III AKI | 3 | 1 | 1 | 1 | 3

4. Secondary Outcome: Duration of AKI
Description: AKI is defined using the Scr-KDIGO criteria. Duration of AKI is defined as the number of days from start of AKI (SCr-KDIGO) where either SCr increase ≥ 0.3 mg/dL above pre-AKI reference point (if the value exists) or if SCr increase ≥1.5 times baseline or dialysis in the first 7 days up to discharge if prior to 7 days.
Time Frame: 7 days OR up to discharge after surgery
Population: Per Protocol Analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | THR-184 Dose 1 | THR-184 Dose 2 | THR-184 Dose 3 | THR-184 Dose 4
Number analyzed (Participants) | 93 | 24 | 29 | 91 | 71
days | 3.7 (2.44) | 2.4 (1.80) | 2.8 (1.92) | 3.4 (2.49) | 3.5 (2.47)

5. Other Pre Specified Outcome: Composite of Death, Dialysis, or Sustained Impaired Renal Function
Description: Sustained impaired renal function defined as a 35% increase in SCr from baseline at Day 30.
Time Frame: Day 30
Population: Per Protocol Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | THR-184 Dose 1 | THR-184 Dose 2 | THR-184 Dose 3 | THR-184 Dose 4
Number analyzed (Participants) | 93 | 24 | 29 | 91 | 71
Participants
  Subjects meeting Endpoint | 11 | 4 | 5 | 11 | 12
  Subjects not meeting Endpoint | 77 | 17 | 20 | 73 | 47
  Subjects excluded from measure | 5 | 3 | 4 | 7 | 12

6. Other Pre Specified Outcome: Composite of Death, Dialysis, or Sustained Impaired Renal Function
Description: Sustained impaired renal function defined as a 35% increase in SCr from baseline at Day 30.
Time Frame: Day 30
Population: Per Protocol Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | THR-184 Dose 1 | THR-184 Dose 2 | THR-184 Dose 3 | THR-184 Dose 4
Number analyzed (Participants) | 93 | 24 | 29 | 91 | 71
Participants
  Subjects meeting Endpoint | 14 | 5 | 4 | 9 | 16
  Subjects not meeting Endpoint | 59 | 13 | 15 | 65 | 55
  Subjects excluded from measure | 20 | 6 | 10 | 17 | 0

ADVERSE EVENTS:
Time Frame: Data were collected over approximately 90 days post-cardiac surgery, with a 14 day Screening Period prior to surgery.
Description: Systematic Assessment: each patient was evaluated at least once a day until day 7 post-surgery or until discharge from the hospital. Subjects returned for a follow-up visit on Day 30 and Day 90 and follow-up phone calls were conducted on Day 14 and Day 60.
Arm/Group | Placebo | THR-184 Dose 1 | THR-184 Dose 2 | THR-184 Dose 3 | THR-184 Dose 4
Serious Adverse Events (participants affected / at risk) | 48/115 | 21/45 | 28/47 | 50/119 | 43/105
Other Adverse Events (participants affected / at risk) | 112/115 | 41/45 | 46/47 | 116/119 | 103/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | THR-184 Dose 1 (N=45) | THR-184 Dose 2 (N=47) | THR-184 Dose 3 (N=119) | THR-184 Dose 4 (N=105)
Atrial fibrillation (Cardiac disorders) | 7 | 0 | 3 | 4 | 3
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 1 | 4 | 1
Cardiac arrest (Cardiac disorders) | 1 | 2 | 2 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Arrythmia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Nodal rhythm (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 5 | 1 | 2 | 3 | 4
Cardiogenic shock (Cardiac disorders) | 4 | 2 | 2 | 2 | 2
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Low cardiac output syndrome (Cardiac disorders) | 2 | 0 | 0 | 0 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 1 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Dressler's syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Myocardial rupture (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Systolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 5 | 6 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 1 | 1 | 1 | 4
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 1 | 2
Sepsis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Diabetic foot infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Wound abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis escherichia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Endocarditis enterococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 0 | 3 | 2 | 1
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Mental status changes postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural stroke (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Wound dishiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Neurological symptom (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Coma (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Stupor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 4 | 4
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 3 | 1 | 1 | 1 | 3
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Haemodynamic instability (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Air embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 2 | 1
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Device malfunction (General disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 1 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Hepatic congestion (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Catatonia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Optic neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Chrondocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Implantable defibrillator replacement (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Wound drainage (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | THR-184 Dose 1 (N=45) | THR-184 Dose 2 (N=47) | THR-184 Dose 3 (N=119) | THR-184 Dose 4 (N=105)
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 6 | 3
Hypokalemia (Metabolism and nutrition disorders) | 24 | 7 | 7 | 35 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 16 | 9 | 10 | 27 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 5 | 4 | 6 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 6 | 5 | 17 | 10
Acid-base disorders (Metabolism and nutrition disorders) | 3 | 2 | 3 | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 2 | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 8 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 6 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 5 | 3 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 7 | 10 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 5 | 4
Procedural pain (Injury, poisoning and procedural complications) | 22 | 9 | 9 | 34 | 27
Anaemia postoperative (Injury, poisoning and procedural complications) | 5 | 6 | 1 | 8 | 5
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 1 | 4 | 3 | 3
Wound complication (Injury, poisoning and procedural complications) | 6 | 4 | 3 | 6 | 7
Anaemia (Blood and lymphatic system disorders) | 34 | 18 | 13 | 31 | 25
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 11 | 9 | 17 | 11
Leukocytosis (Blood and lymphatic system disorders) | 6 | 4 | 3 | 8 | 3
Coagulopathy (Blood and lymphatic system disorders) | 5 | 1 | 3 | 4 | 2
Nausea (Gastrointestinal disorders) | 24 | 14 | 9 | 24 | 25
Vomiting (Gastrointestinal disorders) | 4 | 6 | 4 | 2 | 7
Constipation (Gastrointestinal disorders) | 19 | 10 | 4 | 14 | 11
Oral soft tissue conditions (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0
Hypotension (Vascular disorders) | 25 | 8 | 14 | 21 | 19
Hypertension (Vascular disorders) | 5 | 4 | 6 | 9 | 5
Vascular haemorrhagic disorders (Vascular disorders) | 5 | 2 | 3 | 3 | 3
Oedema peripheral (General disorders) | 20 | 7 | 5 | 14 | 19
Asthenia (General disorders) | 4 | 4 | 1 | 4 | 1
Secretion discharge (General disorders) | 2 | 2 | 3 | 0 | 0
Body temperature conditions (General disorders) | 6 | 2 | 3 | 3 | 2
Urinary tract infection (Infections and infestations) | 13 | 7 | 3 | 8 | 11
Postoperative wound infection (Infections and infestations) | 4 | 3 | 1 | 4 | 12
Pneumonia (Infections and infestations) | 10 | 1 | 2 | 4 | 5
Bacterial infectious disorders (Infections and infestations) | 8 | 5 | 3 | 9 | 5
Haemoglobin decreased (Investigations) | 6 | 1 | 2 | 4 | 11
Urine output decreased (Investigations) | 4 | 0 | 1 | 6 | 2
Blood creatinine increased (Investigations) | 2 | 0 | 3 | 3 | 4
Cardiac and vascular investigations (excl. enzyme tests) (Investigations) | 8 | 2 | 2 | 4 | 8
Hepatobiliary investigations (Investigations) | 3 | 5 | 2 | 7 | 7
Blood magnesium decreased (Investigations) | 8 | 2 | 1 | 3 | 0
Blood calcium decreased (Investigations) | 2 | 3 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 3 | 2 | 3 | 2
Protein and chemistry analyses NEC (Investigations) | 5 | 3 | 1 | 5 | 0
Metabolic, nutritional and blood gas investigations (Investigations) | 2 | 3 | 3 | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 18 | 13 | 6 | 23 | 14
Renal failure (Renal and urinary disorders) | 4 | 2 | 4 | 2 | 5
Urinary retention (Renal and urinary disorders) | 7 | 1 | 0 | 4 | 2
Delirium (Psychiatric disorders) | 9 | 1 | 1 | 4 | 7
Confusional state (Psychiatric disorders) | 5 | 3 | 0 | 3 | 4
Insomnia (Psychiatric disorders) | 4 | 5 | 1 | 3 | 12
Agitation (Psychiatric disorders) | 1 | 3 | 2 | 1 | 3
Hypoaesthesia (Nervous system disorders) | 3 | 1 | 4 | 2 | 1
Central nervous system vascular disorders (Nervous system disorders) | 1 | 5 | 0 | 5 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5 | 1 | 2 | 2
Penile and scrotal disorders (excl. infections and inflammations) (Reproductive system and breast disorders) | 1 | 3 | 0 | 0 | 2
Surgical and medical procedures (Surgical and medical procedures) | 4 | 1 | 4 | 2 | 5
Hepatobiliary disorders (Hepatobiliary disorders) | 3 | 4 | 1 | 3 | 4
Atrioventricular block complete (Cardiac disorders) | 2 | 0 | 1 | 8 | 2
Arrhythmia (Cardiac disorders) | 1 | 4 | 0 | 3 | 3
Ventricular fibrillation (Cardiac disorders) | 1 | 2 | 3 | 3 | 2
Atrioventricular block first degree (Cardiac disorders) | 0 | 3 | 3 | 1 | 2
Low cardiac output syndrome (Cardiac disorders) | 11 | 3 | 3 | 7 | 4
Pericardial disorders (Cardiac disorders) | 6 | 3 | 0 | 7 | 3
Fluid overload (Metabolism and nutrition disorders) | 16 | 12 | 13 | 30 | 18
Hyperkalemia (Metabolism and nutrition disorders) | 8 | 5 | 5 | 7 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 11 | 8 | 15 | 10
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 4 | 7 | 4

LIMITATIONS AND CAVEATS:
A limitation of this analysis was that if a subject left the hospital with AKI, the duration of AKI was automatically assigned as 7 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No